CLINICAL TRIAL: NCT06785701
Title: A Randomized Controlled Trial to Assess the Role of Emergent vs Early Endoscopy in Child B and C Cirrhotic Patients With Acute Variceal Bleed (AVB)-EARLY - AVB.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-AVB-01
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Acute Variceal Bleed
MeSH Terms: interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergent Endoscopy (Experimental): UGIE T1-T4 hrs
  Interventions: Procedure: Upper Gastrointestinal Endoscopy
- Early endoscopy (Active Comparator): UGIE T4-T12 hrs
  Interventions: Procedure: Upper Gastrointestinal Endoscopy

INTERVENTIONS:
Procedure: Upper Gastrointestinal Endoscopy — After Entering to emergency based on time of hemetemsis and based on presentation to ER , patient will be assessed and based on hemodyamic stability patient can be taken Early/Emergent endoscopy.

SUMMARY:
Summary-Variceal bleeding - 70% of all upper gastro-intestinal bleeding episodes in patients with portal hypertension, and they result from esophageal varices (EVs), gastric varices (GVs), or ectopic varices.

Management of Acute variceal bleeding includes endoscopic variceal ligation (EVL) along with vasoactive agents. Inspite of successful hemostasis, this is associated with high variceal rebleeding (VRB) in Child B and C cirrhosis and have higher 6-week mortality rates and liver related adverse events. From time of presentation to emergent endoscopy that is 4 hours can reduce the mortality when compared early endoscopy within 4-12 hours so that mortality rate related to bleed can reduced and early hemostasis can be achieved.

DETAILED DESCRIPTION:
1. Aim and Objectives -To assess the role of Emergent Endoscopy vs Early endoscopy in patients with Acute variceal bleed in CHILD B&C Cirrhosis.
2. Hypothesis - Early use of endoscopy along with adequate resuscitation and medical optimization in patients with Child B/C cirrhosis would lead to higher rates of endoscopic hemostasis thereby associated with better clinical outcomes, in terms of in hospital mortality rate and Liver failure related mortality in post bleed, recurrent bleeding rates.

Study population- Patient presenting with AVB as per definition in Child B &C cirrhotics.

Study design- Randomized Control Trial Non Inferior Trial. Study area- ILBS , Delhi Intervention: Patient after screening for all exclusion criteria will be randomized into either Emergent endoscopy or Early endoscopy

Monitoring and assessment: All patients would undergo vital and baseline parameter screening before randomization. Based on randomization they will undergo the Endoscopy procedure.Post procedure patient will be followed and evaluated for rebleed, mortality, liver related events if any like Hepatic encephalopathy, Ascites, Ischemic hepatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Child B and C cirrhotic patients with history of AVB
2. >18YRS and <75 yrs.
3. Fluid responsive within 1 hour after resuscitation

Exclusion Criteria:

1. EHPVO / NCPH
2. Lack of consent Pregnancy
3. Child A cirrhotics
4. Severe cardiopulmonary disease requiring optimization (Deemed contraindication for endoscopy within 12 hours).
5. Need of Dual vasopressors at presentation In Hospital patients with Bleed
6. HCC patients with AVB
7. Patients presented with AVB on going antiplatelets/anticoagulants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of mortality within 6 weeks in Child B&C | 6 weeks

SECONDARY OUTCOMES:
Proportion of rebleed within 6 weeks in Chid B &C | 6 weeks
Proportion of patients rebleed at D5 | Day 5
Proportion of patients required repeated hospital admissions and number days pf hospitalisation | 6 weeks
Proportion of LRE post bleed within 6 weeks - Ascites/ Hepatic Encephalopathy | 6 weeks
Proportion of patients developing Ischemic hepatitis | 6 weeks
Patients need of TIPS/BRTO/EUS in AVB | 6 weeks
Percentage of endoscopic hemostasis is achieved at 24 hours | 24 hours
Percentage requiring ICU saty and duration of saty post AVB | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided